CLINICAL TRIAL: NCT02767856
Title: Intense vs Standard Regimens of Intermittent Occlusion Therapy for Unilateral Moderate Amblyopia in Children
Brief Title: Regimens of Intermittent Occlusion Therapy for Amblyopia in Children
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI changed the institution.
Sponsor: Salus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HJW1604
Record Dates: First submitted 2016-05-08; First posted 2016-05-10 (Estimated); Results first posted 2022-07-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-05

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intense 12-hour IO-therapy Group (Experimental): Participants wear 12-hour daily IO-therapy glasses for 4 weeks
  Interventions: Device: IO-therapy Glasses
- Standard 4-hour IO-therapy Group (Active Comparator): Participants wear 4-hour daily IO-therapy glasses for 12 weeks
  Interventions: Device: IO-therapy Glasses

INTERVENTIONS:
Device: IO-therapy Glasses

SUMMARY:
This study is designed to answer the question: What if the Intermittent Occlusion (IO-therapy) glasses were prescribed all day (12-hours) in which the total time of treatment only took 4 weeks instead of the current treatment time (4 hours) in which it takes 12 weeks?

Children aged 3- to 8-years with untreated moderate unilateral amblyopia will be enrolled and randomized into 2 groups: 1) Intense 12-hour IO-therapy Group for 4 weeks treatment; or 2) Standard 4-hour IO-therapy glasses Group for 12 weeks treatment.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met for the patient to be enrolled in the study:

1. Age 3 to < 8 years
2. Unilateral amblyopia associated with strabismus (comitant or incomitant), anisometropia, or both

   Criteria for strabismus: At least one of the following criteria must be met:
   * Heterotropia at distance and/or near fixation on examination (with or without spectacles)
   * History of strabismus surgery
   * Documented history of strabismus which is no longer present (which in the judgment of the investigator could have caused amblyopia)

   Criteria for anisometropia: At least one of the following criteria must be met:
   * >0.50 D difference between eyes in spherical equivalent
   * >0.50 D difference between eyes in astigmatism in any meridian
3. Amblyopic eye has no myopia (> -0.25 D spherical equivalent).
4. Visual acuity, measured in each eye without cycloplegia within 7 days prior to enrollment using the ATS single-surround HOTV letter protocol as follows:

   * Visual acuity in the amblyopic eye between 20/40 and 20/80 inclusive
   * Visual acuity in the sound eye 20/32 or better
   * Inter-eye acuity difference ≥ 2 logMAR lines (i.e., amblyopic eye acuity at least 2 lines worse than sound eye acuity)
5. No previous amblyopia treatment within 6 months.
6. Spectacle correction (if applicable) for measurement of enrollment visual acuity must meet the following criteria and be based on a cycloplegic refraction within 6 months:

   * Requirements for spectacle correction:
   * For patients meeting criteria for only strabismus

     * Hypermetropia if corrected must not be undercorrected by more than +1.50 D spherical equivalent, and the reduction in plus sphere must be symmetric in the two eyes. Otherwise, spectacle correction is at investigator discretion.
   * For patients meeting criteria for anisometropia or combined-mechanism

     * Spherical equivalent must be within 0.50 D of fully correcting the anisometropia
     * Hypermetropia must not be undercorrected by more than +1.50 D spherical equivalent, and reduction in plus must be symmetric in the two eyes
     * Cylinder power in both eyes must be within 0.50 D of fully correcting the astigmatism
     * Cylinder axis in the spectacle lenses in both eyes must be within 6 degrees of the axis of the cycloplegic refraction

   Spectacles meeting above criteria must be worn either:
   * for 4 weeks immediately prior to enrollment, or
   * until visual acuity in amblyopic eye is stable (defined as two consecutive visual acuity measurements at least 4 weeks apart with no improvement of one line or more)
   * An acuity measurement done any of the following ways may be considered the first of two consecutive measurements:

     * in current glasses,
     * in trial frames with full correction of hypermetropia with cycloplegia, or
     * in new glasses.
7. Wearing optimal spectacle correction for a minimum of 4 weeks at the time of enrollment.
8. Ocular examination within 6 months prior to enrollment.
9. Gestational age > 34 weeks and birth weight > 1500 grams
10. Parent willing to accept randomization
11. Parent willing to be contacted and has access to phone
12. Parent does not anticipate relocation outside area within study period.

Exclusion Criteria:

1. Amblyopic eye has myopia worse than -3.00 D spherical equivalent.
2. Prior intraocular or refractive surgery
3. Ocular pathologies that impact vision
4. Cognitive impairment that prohibits accurate data collection

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus University, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang J, Malik A, Jin J, Pang Y, Yin K, Allen M, Grigorian A, Scombordi B, Bailey J, Aljohani S, Funari K, Shoge R, Meiyeppen S, Myung J, Soni A, Neely DE. Intense versus standard regimens of intermittent occlusion therapy for unilateral moderate amblyopia in children: study protocol for a randomized controlled trial. Trials. 2020 Apr 28;21(1):361. doi: 10.1186/s13063-020-04284-4. PMID 32345348

RESULTS

PARTICIPANT FLOW:
Groups:
- Intense 12-hour IO-therapy Group: Participants wear 12-hour daily IO-therapy glasses for 4 weeks
  IO-therapy Glasses
- Standard 4-hour IO-therapy Group: Participants wear 4-hour daily IO-therapy glasses for 12 weeks
  IO-therapy Glasses
Period: Overall Study
Arm/Group | Intense 12-hour IO-therapy Group | Standard 4-hour IO-therapy Group
Started | 18 | 14
Completed | 7 | 12
Not Completed | 11 | 2
Not completed — Lost to Follow-up | 9 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intense 12-hour IO-therapy Group | Standard 4-hour IO-therapy Group | Total
Number analyzed (Participants) | 18 | 14 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18 | 14 | 32
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.7 (1.4) | 6.0 (1.5) | 5.8 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 6 | 17
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 14 | 8 | 22
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 14 | 10 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Visual acuity at baseline [Mean (Standard Deviation); unit: logMAR] | 0.38 (0.11) | 0.385 (0.11) | 0.38 (0.11)

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity Improvement
Description: visual acuity difference between the primary outcome measure and baseline in the amblyopic eye; visual acuity was measured with ATS- HOTV method
Time Frame: 4 weeks for the Intense Group and 12 weeks for the Standard Group
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Intense 12-hour IO-therapy Group | Standard 4-hour IO-therapy Group
Number analyzed (Participants) | 7 | 12
logMAR | 0.17 (0.11) | 0.13 (0.12)
Statistical Analysis 1: Comparison: Intense 12-hour IO-therapy Group vs Standard 4-hour IO-therapy Group; Baseline and primary visit outcome; Test type: Equivalence — The study did not enroll enough samples. The stats here are only for reference; p = 0.48, t-test, 2 sided; Mean Difference (Net) = 0.04, 95% CI 2-sided [-0.08 to 0.16]

2. Secondary Outcome: Stereoacuity Test
Description: Stereoacuity in arcsec was converted to log scale. so log10(stereo) will be reported.
  The higher value indicates a poorer binocular visual function.
Time Frame: 4 weeks for the Intense Group and 12 weeks for the Standard Group
Measure: Mean (Standard Deviation); unit: log(arcsec)
Arm/Group | Intense 12-hour IO-therapy Group | Standard 4-hour IO-therapy Group
Number analyzed (Participants) | 7 | 11
log(arcsec) | 3.04 (0.78) | 3.16 (0.93)
Statistical Analysis 1: Comparison: Intense 12-hour IO-therapy Group vs Standard 4-hour IO-therapy Group; Test type: Equivalence — The study did not reach the target sample size. the stats are for reference; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [-0.75 to 0.99]

3. Secondary Outcome: Objective Total Treatment Hours
Description: Objective total treatment hours at the primary outcome visit measured with a microsensor
Time Frame: 4 weeks for the Intense Group and 12 weeks for the Standard Group
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Intense 12-hour IO-therapy Group | Standard 4-hour IO-therapy Group
Number analyzed (Participants) | 6 | 10
hour | 135.5 (30.5) | 109.2 (58.7)
Statistical Analysis 1: Comparison: Intense 12-hour IO-therapy Group vs Standard 4-hour IO-therapy Group; Test type: Equivalence — The study did not reach the target sample size. The stats are for reference; p = 0.26, t-test, 2 sided; Mean Difference (Final Values) = 26.3, 95% CI 2-sided [-21.75 to 74.20]

4. Secondary Outcome: Objective Adherence
Description: objective adherence measured with a microsensor to the treatment regimen
Time Frame: 4 weeks for the Intense Group and 12 weeks for the Standard Group
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Intense 12-hour IO-therapy Group | Standard 4-hour IO-therapy Group
Number analyzed (Participants) | 6 | 10
percent | 43.0 (12.7) | 54.1 (40.6)
Statistical Analysis 1: Comparison: Intense 12-hour IO-therapy Group vs Standard 4-hour IO-therapy Group; Test type: Equivalence — The study did not reach the target sample size. The stats are for reference; p = 0.44, t-test, 2 sided; Mean Difference (Final Values) = 11.1, 95% CI 2-sided [-41.3 to 19.3]

ADVERSE EVENTS:
Time Frame: From enrollment until the primary outcome visit and the follow-up visits. For the Intense Group, the primary outcome visit is at 4 weeks, and they also follow up at 12 weeks; for the Standard group, the primary outcome visit is at 12 weeks, if improved, they follow up at 24 weeks.
Description: Reverse amblyopia: defined as two or more logMAR lines worse in the fellow non-amblyopic eye at the primary visit; significant changes in ocular alignment: defined as deviation changes of ≥10Δ; any injury associated with IO-therapy glasses or the microsensor.
Arm/Group | Intense 12-hour IO-therapy Group | Standard 4-hour IO-therapy Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/12
Other Adverse Events (participants affected / at risk) | 0/7 | 0/12

LIMITATIONS AND CAVEATS:
Termination leads to small numbers of subjects analyzed. Several participants lost follow-up. One patient withdrew from the study due to a dislike of the device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/56/NCT02767856/Prot_SAP_ICF_000.pdf